CLINICAL TRIAL: NCT05872711
Title: Low Carbohydrate Versus Mediterranean Diet in Adolescents With Type 1 Diabetes: A Randomized Control Trial
Brief Title: Low Carbohydrate Versus Mediterranean Diet in Adolescents With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Orit Hamiel, Head of Pediatric Endocrinology Department in Sheba Medical Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SHEBA-18-5537-OH-CTIL
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
Keywords: Adolescents; Glycemic targets; Low carbohydrate diet; Mediterranean diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: The study design is a randomized, parallel assignment clinical trial without blinding (open label) due to the impracticality of blinding diets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet (Experimental): The LCD will provide 50-80g of carbohydrate per day with no caloric restriction. The planned macronutrient compositions (percentages of the total calories) of the diet were: 15-20% carbohydrate (<80 g/day), 33% protein and 58% total fat.
  Interventions: Other: Low carbohydrate diet
- Mediterranean diet (Active Comparator): The MED group was prescribed a moderate-fat MED, rich in vegetables and low in red meat, with poultry and fish preferred to beef and lamb. The primary sources of added fat were 30 to 45 g of olive oil and a handful of nuts (five to seven nuts <20g) per day. The planned macronutrient compositions of the diet were 40-50% carbohydrate, 25% protein and 35% total fat. The diet is based on the recommendations of Willett and Skerrett
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet — In order to maintain equal intensity of treatment, each patient will get a cooking workshop and received a personalized diet regime at baseline, based on the randomly assigned diet. Format and quality of the materials are similar.
  All diet plans are individualized and matched for energy intake personally . Participants will meet individually with the dietitian for diet instruction and support at week 1,2,4,7,10,12 and thereafter at 24 weeks for a total of seven frontal meetings. Twice during the first 12 weeks the dietician will conduct 10-15-minute motivational telephone calls with all the participants.

SUMMARY:
The goal of this clinical trial is to compare the effect of low carbohydrate diet versus Mediterranean diet on blood sugar values in adolescents with type 1 diabetes.

The main question aims to answer whether a low carbohydrate diet is as effective as the Mediterranean diet for better glycaemic control in type 1 adolescents.

The investigators are also aiming to check whether low carbohydrate diet is safe and does not elevate cholesterol blood levels and whether the diet is adherable among youth with type 1 diabetes.

Participants with type 1 diabetes wearing a continuous glucose monitor and that will sign an informed consent will be randomly selected for 2 groups. One group will get the Mediterranean diet program and the other will get the low carbohydrate diet program, both for a duration of six months. Each participant will attend a cooking workshop at the beginning of the study. Blood work and stool samples will be taken at the beginning and 3 times through the study periodd. Each participant will attend meetings with the dietician thorough the period of the study.

DETAILED DESCRIPTION:
Background and objective: Improved glycemic control of type 1 diabetes (T1DM), with low rates of adverse events was reported via an online community of children and adults who consume a of low carbohydrate diet (LCD). The investigators aim to compare the effects of a low carbohydrate diet (LCD) with those of a Mediterranean diet on glycemic control, lipid profile, bone metabolites and the microbiome profile in adolescents with type 1 diabetes.

Design A randomized, controlled trail. Families of adolescents in the Diabetes clinic in Edmond and Lily Safra Children's Hospital will be approached and offered to participate in a dietary intervention study. After participants will sign the informed consent, they will randomly be assigned into 2 diet treatment groups, the LCD (n=20) and the Mediterranean diet (n=20). Baseline nutrition teaching session and training and will be conducted for all participants and their parents. Participants will attend visit with the dietician at baseline, 2, 4, 8,12 weeks and will be given a 3-day food dairy to complete twice in that period. Measurements of weight, height, blood pressure, HbA1c, Time in range, number of hypoglycemia, lipid profile, creatinine, bone metabolites will be measured at baseline and 12 and 24 weeks and gut bacteria profile at baseline and at 24 weeks. Personality, quality of life, and socioeconomic questionnaires will be given to children and their parents.

Contribution of the suggested research:

In this research the investigators are aiming to show that LCD is as good as Mediterranean diet with improved glycemic control, safe, and adherable for adolescent with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Connected to a continuous glucose monitoring (CGM)

Exclusion Criteria:

* History of eating disorder
* Family history of mental disorders

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of time in range (TIR) 70-180 mg/dl after following a LCD or a MD in adolescents with T1DM. | The change of TIR between baseline and after six months
  Time spent in range (TIR) 70-180 mg/dl assessed by CGM was downloaded at each visit with the dietician. Severe hypoglycemia was defined as an episode requiring assistance and was confirmed by documentation of a blood glucose value less than 54 mg per deciliter

SECONDARY OUTCOMES:
Evaluation of the influence of LCD vs. MD on HbA1c. | The change between baseline and after six months
  Blood test for Hba1c will be taken at baseline and 24 weeks. Insulin dose and glycemic variability will be taken at each visit with the dietician from=n the pump and sensor downloads.
Assessment of the impact of dietary changes after an LCD vs. MD on gut dysbiosis | The change between baseline and after six months
  Three stool samples will be take from each participant, and kept in -80c until being investigated in a lab
Assessment of the impact of both diets on bone turnover measures. | The change of bone turnover at baseline and after six months
  Blood samples will be taken from the participants after a 12-hr fast at baseline,12 and 24 weeks. Bone markers: procollagen type 1 amino-terminal propeptide (P1NP) and bone resorption C-terminal telopeptide of type 1 collagen (CTx1) as well as cholesterol, LDL cholesterol, triglyceride and HDL cholesterol.
Assessment of the impact of dietary changes after an LCD vs. MD on quality of life. | The change between baseline and after six months in the quality of life.
  Quality of life questionnaire for type 1 diabetes adolescents will be given at baseline and after 6 months. A higher score reflects a better equality of life.
Change in BMI after LCD vs. MD | BMI change at baseline and after six months
  Measured height and weight will be taken at baseline and after 6 months of intervention in both arms and will be calculated into BMI. The outcome is the change in BMI at baseline and at the end of the intervention.
Change in diet LCD vs. MED | Baseline and after six months
  FFQ (food frequency questionnaire) will be given at baseline and after 6 months to both arms, change of micronutrients and macronutrients will be calculated according to the questionnaire
Change in LDL cholesterol | Baseline and after 6 months
  Blood test will be taken at baseline and after six months of intervention. Change in LDL cholesterol before and after the diets.

CONTACTS AND LOCATIONS:
Overall Officials: Orit Pinhas-Hamiel, MD, Principal Investigator — Head oh Pediatric Endocrinology Unit
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lennerz BS, Barton A, Bernstein RK, Dikeman RD, Diulus C, Hallberg S, Rhodes ET, Ebbeling CB, Westman EC, Yancy WS Jr, Ludwig DS. Management of Type 1 Diabetes With a Very Low-Carbohydrate Diet. Pediatrics. 2018 Jun;141(6):e20173349. doi: 10.1542/peds.2017-3349. Epub 2018 May 7. PMID 29735574
- [Result] Schmidt S, Christensen MB, Serifovski N, Damm-Frydenberg C, Jensen JB, Floyel T, Storling J, Ranjan A, Norgaard K. Low versus high carbohydrate diet in type 1 diabetes: A 12-week randomized open-label crossover study. Diabetes Obes Metab. 2019 Jul;21(7):1680-1688. doi: 10.1111/dom.13725. Epub 2019 Apr 21. PMID 30924570

DOCUMENTS (1):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT05872711/Prot_000.pdf